CLINICAL TRIAL: NCT00171158
Title: An Extension to a Phase II Open-label Study to Determine the Safety and Anti-leukemic Effects of STI571 in Patients With Philadelphia Chromosome-positive Chronic Myeloid Leukemia in Myeloid Blast Crisis
Brief Title: An Extension Study of the Safety and Anti-leukemic Effects of Imatinib Mesylate in Participants With Philadelphia Chromosome-positive Chronic Myeloid Leukemia in Blast Crisis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A0102E2; 2005-001380-61 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Philadelphia Chromosome Positive CML
Keywords: Chronic Myelogenous Leukemia; CML; Philadelphia Chromosome; Blast crisis; Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Blast Crisis | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib Mesylate (STI571) (Experimental): Participants initially received STI571 capsules or tablets, orally, initially once daily (400 mg) or (600 mg). The dosage was escalated from 400 mg to 600 mg and from 600 mg to 800 mg, on an individual basis as per the investigator's judgement. Treatment continued until death, or the development of intolerable toxicity, or the participant was considered not to benefit from treatment, whichever came first.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: Gleevec/Glivec

SUMMARY:
This extension II study allowed for further follow-up of the disease under treatment with imatinib mesylate and allow the participants to continue to receive imatinib mesylate.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Philadelphia chromosome positive chronic myelogenous leukemia (CML) in myeloid blast crisis (including both newly diagnosed and the participants who received prior therapy for accelerated or blastic phases), defined as either:

1. ≥ 30% blast in peripheral blood and /or bone marrow
2. by flow cytometry criteria

2. To be categorized as "newly diagnosed", participants with CML in blast crisis were not to have received specific therapy for CML accelerated or blast phases, with the exception of interferon-alpha or hydroxyurea.

3. serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) not more than 3 times the upper limit of the normal range (ULN) (or not more than 5 times the ULN if clinically suspected leukemic involvement of the liver), serum creatinine concentration not more than 2 times the ULN, and total serum bilirubin level not more than 3 times the ULN at the laboratory where the analyses were performed.

4. A negative pregnancy test in participants of childbearing potential.

Exclusion Criteria:

1. Participants with an eastern cooperative oncology group (ECOG) performance status score ≥ 3.
2. Participants previously treated for blast crisis were not to have received any of the following with respect to Day 1 of the study: busulfan within six weeks, interferon-alpha within 48-hours, hydroxyurea within 24-hours, homoharringtonine within 14 days, low-dose, moderate dose or high dose cytosine arabinoside within 7, 14 and 28 days respectively, anthracyclines, mitoxantrone, or etoposide within 21 days.
3. Participants receiving any hematopoietic stem cell transplantation within six weeks of Day 1.
4. Participants receiving any other investigational agents within 28 days of Day 1.
5. Participants with Grade 3/4 cardiac disease or any other serious concurrent medical conditions.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1999-07-26 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Dana Faber Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Poitiers, France
- Germany (4):
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
- Italy (2):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Monza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The overall study was conducted at 28 investigative sites in 6 countries from 26 July 1999 to 22 April 2013. A total of 260 participants were enrolled in the core Study CSTI57A0102, of which 21 participants completed the treatment and were enrolled in the extension Study CSTI571A0102E1. 13 participants discontinued from the extension Study CSTI571A0102E1, and 8 of them were enrolled in the extension Study CSTI571A0102E2.
Pre-assignment Details: The study enrolled 8 participants with myeloid blast crisis who completed their participation in Study CSTI571A0102E1.
Groups:
- Imatinib Mesylate (STI571): Participants initially received STI571 capsules or tablets, orally, initially once daily (400 mg) or (600 mg). The dosage was escalated from 400 mg to 600 mg and from 600 mg to 800 mg on an individual basis as per the investigator's judgement. Treatment continued until death, or the development of intolerable toxicity, or the participant was considered not to benefit from treatment, whichever came first.
Period: Core Study
Arm/Group | Imatinib Mesylate (STI571)
Started | 260
Completed | 21
Not Completed | 239
Not completed — Death | 27
Not completed — Unsatisfactory therapeutic effect | 163
Not completed — Protocol Violation | 4
Not completed — Administrative problems | 1
Not completed — Adverse event, non-fatal | 21
Not completed — Consent withdrawn by subject | 6
Not completed — No longer required drug (BMT) | 14
Not completed — Abnormal Laboratory Values | 2
Not completed — Lost to Follow-up | 1
Period: E2 Extension
Arm/Group | Imatinib Mesylate (STI571)
Started (Participants that completed the core study entered the Extension 1 (E1) of the study, of which 13 participants discontinued the study. 8 participants entered Extension (E2).) | 8
Completed | 1
Not Completed | 7
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all participants who enrolled in the study.
Arm/Group | Imatinib Mesylate (STI571)
Number analyzed (Participants) | 260
Age, Continuous [Median (Full Range); unit: years] | 56 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 136

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the number of events of death, expressed as a percentage, from the start of treatment to death, due to any reason.
Time Frame: From first dose until death of the patient, up to 14 years.
Population: The Intent-to-treat (ITT) population included all participants who enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib Mesylate (STI571)
Number analyzed (Participants) | 260
percentage of participants | 89.2

2. Primary Outcome: Overall Survival (by Month)
Description: Overall survival was defined as the time between start of treatment and death due to any reason. Overall survival for the participants was calculated by Kaplan-Meier estimates per month. The time was censored at the date of last contact for participants who discontinued treatment and were in survival follow-up.
Time Frame: From first dose until death of the patient, up to 14 years.
Population: The Intent-to-treat (ITT) population included all participants who enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate (STI571)
Number analyzed (Participants) | 260
percentage of participants
  12 Months | 32.7 [27.0 to 38.5]
  24 Months | 18.7 [14.2 to 23.8]
  36 Months | 15.4 [11.2 to 20.2]
  48 Months | 14.5 [10.4 to 19.2]
  60 Months | 9.1 [5.7 to 13.4]
  72 Months | 8.4 [5.2 to 12.7]
  84 Months | 7.5 [4.3 to 11.8]
  96 Months | 7.5 [4.3 to 11.8]
  108 Months | 7.5 [4.3 to 11.8]
  120 Months | 6.6 [3.5 to 11.0]
  132 Months | 5.5 [2.6 to 10.0]
  144 Months | 5.5 [2.6 to 10.0]
  156 Months | 5.5 [2.6 to 10.0]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to 14 years.
Description: After 31 July 2002 no safety data was collected in the clinical database and serious adverse events (SAEs) were reported in the safety database. No drug-related SAEs leading to discontinuation or drug-related deaths were reported after 31 July 2002 in the safety database.
Arm/Group | Imatinib Mesylate (STI571)
Serious Adverse Events (participants affected / at risk) | 0/260
Other Adverse Events (participants affected / at risk) | 0/260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.